CLINICAL TRIAL: NCT02070458
Title: A Phase 1 Study of MLN9708 in Combination With MEC (Mitoxantrone, Etoposide, and Intermediate-Dose Cytarabine) for Relapsed/ Refractory Acute Myelogenous Leukemia (AML)
Brief Title: Ixazomib, Mitoxantrone Hydrochloride, Etoposide, and Intermediate-Dose Cytarabine in Relapsed or Refractory Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE7913; NCI-2014-00371 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); X16014_MLN9708; CASE7913 (Other: Case Comprehensive Cancer Center); P30CA043703 (NIH)
Record Dates: First submitted 2014-02-21; First posted 2014-02-25 (Estimated); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Recurrent Adult Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — ixazomib; Mitoxantrone; Etoposide; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (ixazomib, MEC) (Experimental): Patients receive ixazomib PO on days 1, 4, 8, and 11; they receive mitoxantrone hydrochloride IV, etoposide IV over 1 hour; the receive intermediate-dose cytarabine IV over 6 hours on days 1-6.
  Interventions: Drug: ixazomib; Drug: mitoxantrone hydrochloride; Drug: etoposide; Drug: cytarabine

INTERVENTIONS:
Drug: ixazomib — Given PO
  Other Names: MLN9708; proteasome inhibitor MLN9708
Drug: mitoxantrone hydrochloride — Given IV
  Other Names: CL 232315; DHAD; DHAQ; Novantrone
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213
Drug: cytarabine — Given IV
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside

SUMMARY:
This phase I trial studies the side effects and best dose of ixazomib when given in combination with mitoxantrone hydrochloride, etoposide, and intermediate-dose cytarabine in treating patients with acute myeloid leukemia that is unresponsive to initial induction chemotherapy or recurs following an initial complete remission. Acute myeloid leukemia is a cancer of the bone marrow cells; bone marrow is where blood cells are normally made. Ixazomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as mitoxantrone hydrochloride, etoposide, and intermediate-dose cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Mitoxantrone hydrochloride, etoposide, and intermediate-dose cytarabine are standard treatment for relapsed or refractory acute myeloid leukemia. Giving ixazomib with mitoxantrone hydrochloride, etoposide, and intermediate-dose cytarabine may improve the effectiveness of the chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the dose-limiting toxicities (DLT), maximum tolerated dose (MTD), and the recommended Phase 2 dose of MLN9708 (ixazomib) in combination with mitoxantrone hydrochloride, etoposide, intermediate-dose cytarabine (MEC) in patients with relapsed/ refractory acute myeloid leukemia (AML).

SECONDARY OBJECTIVES:

I. To describe the non-dose limiting toxicities associated with MLN9708 in combination with MEC in patients with relapsed/ refractory AML.

II. To describe any preliminary evidence of clinical activity of this combination (compete response [CR] rate) in relapsed/ refractory AML.

III. To determine the median cluster of differentiation (CD)74 antigen expression in patients achieving a response versus those patients not achieving a response.

IV. To determine if gene expression profile pre- and post-treatment correlates with response to therapy.

OUTLINE: This is a dose-escalation study of ixazomib.

Patients receive ixazomib orally (PO) on days 1, 4, 8, and 11, mitoxantrone hydrochloride intravenously (IV), etoposide IV over 1 hour, and intermediate-dose cytarabine IV over 6 hours on days 1-6.

After completion of study treatment, patients are followed up for 4-5 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care
* Female patients who:

  * Are postmenopausal for at least 1 year before the screening visit, OR
  * Are surgically sterile, OR
  * If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of study drug, AND
  * Must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject (periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception)
* Male patients, even if surgically sterilized (i.e., status post-vasectomy), must agree to one of the following:

  * Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, OR
  * Must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject (periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception)
* Subjects with a prior diagnosis of AML (excluding acute promyelocytic leukemia) based on World Health Organization Classification who did not achieve complete response (CR) with their previous therapy or who have relapsed after achieving a complete response (CR) are eligible; any number of relapses will be eligible.
* Patients must have > 5% blasts in the bone marrow at the time of study enrollment
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, 2, or 3
* Total bilirubin ≤ 1.5 x the upper limit of the normal range (ULN) within 14 days of enrollment
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x ULN within 14 days of enrollment
* Calculated creatinine clearance ≥ 30 mL/min within 14 days of enrollment
* Patients with secondary AML, and patients with a prior autologous and allogeneic bone marrow transplant are eligible
* Patients with an allogeneic transplant must meet the following conditions: the transplant must have been performed more than 90 days before registration to this study, the patient must not have ≥ grade 2 acute graft versus host disease (GvHD) or either moderate or severe limited chronic GvHD, or extensive chronic GvHD of any severity; the patient must be off all immunosuppression for at least 2 weeks
* Echocardiogram or multi gated acquisition (MUGA) scan demonstrating an ejection fraction ≥ 45%

Exclusion Criteria:

* Female patients who are lactating or have a positive serum pregnancy test during the screening period
* Failure to have fully recovered (i.e., ≤ grade 1 toxicity) from the reversible effects of prior chemotherapy, excluding alopecia
* Major surgery within 14 days before enrollment
* Radiotherapy within 14 days before enrollment; if the involved field is small, 7 days will be considered a sufficient interval between treatment and administration of the MLN9708
* Central nervous system involvement; a lumbar puncture does not need to be performed unless there is clinical suspicion of leptomeningeal disease
* Uncontrolled infections
* Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months
* Systemic treatment, within 3 days before the first dose of MLN9708, with strong inhibitors of cytochrome P450, family 1, subfamily A, polypeptide 2 (CYP1A2) (fluvoxamine, enoxacin, ciprofloxacin), strong inhibitors of cytochrome P450, family 3, subfamily A (CYP3A) (clarithromycin, telithromycin, itraconazole, voriconazole, ketoconazole, nefazodone, posaconazole) or strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of Ginkgo biloba or St. John's wort
* Ongoing or active hepatitis B or C virus infection, or known human immunodeficiency virus (HIV) positive
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol
* Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent
* Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of MLN9708 including difficulty swallowing
* Patients with prior malignancy are eligible; however, the patient must be in remission from the prior malignancy and have completed all chemotherapy and radiotherapy at least 6 months prior to registration and all treatment-related toxicities must have resolved; patients with basal cell or squamous cell carcinoma of the skin are eligible regardless of disease status
* Patient has ≥ grade 2 peripheral neuropathy within 14 days of trial enrollment
* Participation in other clinical trials, including those with other investigational agents not included in this trial, within 14 days of the start of this trial and throughout the duration of this trial
* Any standard therapy for leukemia within 14 days before enrollment (except for hydrea)
* Patients who have received prior pulmonary radiation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-10-08 (Actual); Primary Completion 2017-03-17 (Actual); Study Completion 2017-08-15 (Actual)

PRIMARY OUTCOMES:
DLT assessed using the National Cancer Institute (NCI) Common Toxicity Criteria (CTC) scale version 4.03 | Up to 5 weeks
MTD of ixazomib in combination with MEC based on the occurrence of DLT assessed using NCI CTC scale version 4.03 | Up to 5 weeks
Recommended Phase 2 dose | Up to 5 weeks

SECONDARY OUTCOMES:
Incidence of non-DLT assessed using NCI CTC scale version 4.03 | Up to 5 weeks
Complete response (CR) rate | Up to 5 weeks
  The CR rate in this population will be evaluated and explored in a preliminary manner given the small number of patients and different dose levels. The Cheson criteria will be used to analyze response.
Complete remission with incomplete platelet recovery (CRp) rate | Up to 5 weeks
  The CRp rate in this population will be evaluated and explored in a preliminary manner given the small number of patients and different dose levels. The Cheson criteria will be used to analyze response.
Gene expression profile analysis | Up to 5 weeks
  Gene expression profiles will be summarized and compared in patients with response (CR/ CRp) versus patients with no response (all others).
CD74 antigen expression expression analysis | Up to 5 weeks
  The CD74 antigen expression will be summarized and compared in patients with response (CR/ CRp) versus patients with no response (all others).

CONTACTS AND LOCATIONS:
Overall Officials: Anjali Advani, Principal Investigator — Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio
  - University Hospitals Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio